CLINICAL TRIAL: NCT02767076
Title: Paramedian Spinal Anaesthesia for Orthopaedic Knee Surgery: Comparison Between Conventional Blind Land-mark Guided Technique and Real-time Ultrasound Guided Technique: a Randomized Controlled Trial.
Brief Title: Paramedian Spinal Anaesthesia : Comparison Between Land-mark Guided Technique and Real-time Ultrasound Guided Technique.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sohib Mohamed Galal Abdelfatah, anesthesia specialist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: N-15-2016
Record Dates: First submitted 2016-04-22; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Paramedian Spinal Anaesthesia; Real Time Ultrasound Guiding
Keywords: paramedian spinal anesthesia; real time; ultrasound; knee surgeries; conventional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional (Active Comparator): conventional paramedian spinal anesthesia
  Interventions: Procedure: conventional paramedian spinal anesthesia
- Ultrasound (Experimental): ultrasound guided paramedian spinal anesthesia
  Interventions: Device: ultrasound guided paramedian spinal anesthesia

INTERVENTIONS:
Procedure: conventional paramedian spinal anesthesia — land mark guided paramedian spinal anesthesia
  Arms: Conventional
Device: ultrasound guided paramedian spinal anesthesia — real time ultrasound guided paramedian spinal anesthesia
  Arms: Ultrasound

SUMMARY:
To identify the value of using the ultrasound in applying a commonly used regional anaesthetic procedure (spinal anaesthesia) when compared with the conventional landmark guided approach, regarding the efficiency of the anaesthetic technique, incidence of associated common complications and patient's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I-II patients
2. Patient's consented approval
3. Males or Females
4. Aged 18-60 years old
5. Body mass index less than 30
6. Scheduled for orthopaedic knee surgeries

Exclusion Criteria:

1. Age less than 18, and more than 60 years
2. Body mass index more than 30
3. Patient refusal or failure to obtain consent
4. Patient in whom spinal anaesthesia is contraindicated (infection at the site of needle insertion, coagulopathy reflected by values of INR≥ 1.2 or platelets count≤ 75.000, or receiving oral anticoagulants)
5. Known sensitivity to local anaesthetics
6. Pre-existing neurological disorder or neuromuscular disease
7. Clinically obvious or known spinal deformity or previous spinal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Number of puncture attempts | during the time taken for introducing the regional anesthetic technique in the intraoperative period

SECONDARY OUTCOMES:
Landmark palpation easiness score | during the time taken for introducing the regional anesthetic technique in the intraoperative period
The visibility of the ligamentum flavum-dura mater complex by the US. | during the time taken for introducing the regional anesthetic technique in the intraoperative period
Duration of the anaesthetic procedure | during the time taken for introducing the regional anesthetic technique in the intraoperative period
The incidence of paraesthesia and backache | during the time taken for introducing the regional anesthetic technique in the intraoperative period
The incidence of failure of introducing spinal anaesthesia using each of the study techniques. | during the time taken for introducing the regional anesthetic technique in the intraoperative period
Patient's satisfaction score regarding the anaesthetic technique | within 2 hours in the postoperative period
Post dural puncture headache (incidence-onset-duration-severity) | within 3 days after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo, Cairo Governorate, Egypt